CLINICAL TRIAL: NCT02992223
Title: Retrospective Collection of Data on Patient With Relapsed/Refractory Aggressive Non Hodgkin Lymphoma Treated With Y90 Ibritumomab Tiuxetan Radioimmunotherapy Plus High-Dose Chemotherapy and Autologous Stem Cell Transplant
Brief Title: Retrospective Analysis on Relapsed/Refractory Aggressive Non Hodgkin Lymphoma Treated With Z-BEAM Plus ASCT
Status: Completed | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Barbara Botto, MD, A.O.U. Città della Salute e della Scienza
Other Study IDs: Oss_Z-BEAM
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Refractory B-Cell Non-Hodgkin Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma
Keywords: Aggressive B-cell non-Hodgkin Lymphoma; Relapsed; Refractory; Zevalin; Y90 Ibritumomab Tiuxetan; Autologous stem cell transplant; BEAM; Recurrent
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluate if Y90 Ibritumomab Tiuxetan Radioimmunotherapy in addition to standard high dose chemotherapy followed by autologous stem cell transplant could improve prognosis in patients affected by relapsed/refractory aggressive non Hodgkin lymphoma

ELIGIBILITY:
Inclusion Criteria:

* High Risk Relapsed/refractory aggressive non-hodgkin lymphoma defined as:
* Progressive disease
* Early relapse (within 12 months from response)
* Recurrent relapse
* Treated with salvage chemotherapy followed by Y90 Ibritumomab Tiuxetan plus high-dose chemotherapy and Autologous stem cell transplant
* Age > 18 years
* Previous treatment with Rituximab
* Written informed consent

Exclusion Criteria:

* Patient with no complete data available for collection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient With Relapsed/Refractory Aggressive Non Hodgkin Lymphoma treated with Y90 Ibritumomab Tiuxetan Radioimmunotherapy Plus High-Dose Chemotherapy and Autologous Stem Cell Transplant
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Date of last follow-up for at least 18 months (up to 78 months)
  Time to last follow-up or death
Progression Free Survival | From first response to last follow-up for at least 18 month (up to 78 months)
  Time from last response to nearest relapse or follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Botto, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza

IPD SHARING:
Plan to Share IPD: Yes
paper publication